CLINICAL TRIAL: NCT01267851
Title: A Large Multicentre Clinical Database and Biobank of Patients With Gynecologic Neoplasms
Brief Title: Clinical Database and Biobank of Patients With Gynecologic Neoplasms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Zhejiang University (Other); Hunan Province Tumor Hospital (Other); Guangxi Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); West China Second University Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Shanghai First Maternity and Infant Hospital (Other); Peking University People's Hospital (Other); Wuhan Central Hospital (Other)
Responsible Party: Principal Investigator, Ding Ma, Director of the department of Obstetrics and Gynecology, Tongji Hospital, Huazhong University of Science and Technology
Other Study IDs: GM2010-06-02
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Cervical Cancer; Ovarian Cancer; Endometrial Cancer; Choriocarcinoma; Uterine Myoma; Endometriosis
Keywords: gynecologic disease
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Choriocarcinoma; Myofibroma; Endometriosis; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The database and biobank establishment started in 1997 in our institute. However, the sample size was too small with respect to our clinical and fundamental scientific research's requirement. Thus the Chinese gynecological oncology study (GOS) group was established to create a large multicentre database and biobank of patients with gynecologic diseases.

DETAILED DESCRIPTION:
The database contains clinical and epidemiologic information about patients with gynecologic neoplasms, such as cervical carcinoma, ovarian carcinoma, etc. With the data gathered from this database, the investigators could further demonstrate the etiology, risk factor, clinical treatment, and other aspects of the complicated gynecologic diseases. The cervical cancer database v1.10 including more than 10,000 cases and more than 200 variables has been established.

The biobank collects blood, fluids, tissue samples, and related clinical data from consenting patients with gynecologic neoplasms, such as cervical cancer, ovarian cancer, endometrial cancer, choriocarcinoma, uterine myoma, endometriosis. Besides, blood samples of population-based healthy people with informed consent are also collected.

ELIGIBILITY:
Inclusion Criteria:

* patients with informed consent;
* patients with gynecologic diseases;
* patients with intact clinical and pathological information

Exclusion Criteria:

* not included in the inclusion criteria

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: gynecologic diseases, such as cervical cancer, ovarian cancer, endometrial cancer, choriocarcinoma, uterine myoma, endometriosis, as well as part of population-based healthy women
Sampling Method: Probability Sample
Enrollment: 1600000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of HUST, Wuhan, Hubei, China

REFERENCES:
- [Derived] Hu T, Li S, Chen Y, Shen J, Li X, Huang K, Yang R, Wu L, Chen Z, Jia Y, Wang S, Cheng X, Han X, Lin Z, Xing H, Qu P, Cai H, Song X, Tian X, Xu H, Xu J, Zhang Q, Xi L, Deng D, Wang H, Wang S, Lv W, Wang C, Xie X, Ma D. Matched-case comparison of neoadjuvant chemotherapy in patients with FIGO stage IB1-IIB cervical cancer to establish selection criteria. Eur J Cancer. 2012 Oct;48(15):2353-60. doi: 10.1016/j.ejca.2012.03.015. Epub 2012 Apr 13. PMID 22503395